CLINICAL TRIAL: NCT06740708
Title: Scaling Up Community-based Noncommunicable Disease Research Into Practice in Pokhara Metropolitan City of Nepal
Acronym: SCALE NCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB00030203; R01HL172271 (NIH)
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus (T2DM); Tobacco Smoking
Keywords: hypertension; type 2 diabetes mellitus; tobacco smoking; task-sharing; task-shifting; community health workers; female community health volunteers
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCALE-NCD (Intervention) (Experimental): Intervention arm will receive the following two components of the SCALE-NCD intervention package:
  1. FCHV home visits every three months, including measurements, counseling and referral;
  2. Mobile phone messages, including lifestyle modification
  Interventions: Behavioral: SCALE-NCD
- Control (No Intervention): Control arm will receive the usual care in Pokhara Metropolitan City in Nepal.

INTERVENTIONS:
Behavioral: SCALE-NCD — 1. FCHV home visits every three months, including
     * For hypertension i. Blood pressure measurement with digital BP devices ii. Lifestyle counseling iii. Referral if uncontrolled BP (≥140/90 mmHg) for 3 months
     * For type 2 diabetes i. Fasting blood glucose measurement with glucometer ii. Lifestyle counseling focusing on diabetes management iii. Referral if uncontrolled diabetes (≥126mg/dl) for 3 months
     * For current smokers i. Smoking cessation counseling ii. Referral for nicotine replacement therapy if request by participants
  2. Mobile phone messages, including
     * Lifestyle modification
     * Conveyed as voice or text messages, depending on participant preference
  Arms: SCALE-NCD (Intervention)

SUMMARY:
The goal of this clinical trial is to evaluate whether a multifaceted community-based intervention, comprising 1) screening and lifestyle counseling by female community health volunteers (FCHVs); community health workers in Nepal, through home visits, and 2) regular Short Message Service (SMS) messages, can effectively reduce systolic blood pressure (SBP), lower fasting blood glucose, and increase smoking cessation rates among adults living in Pokhara with hypertension, type 2 diabetes, and smoking habits, respectively.

The main research questions are:

* Can FCHV home visits combined with regular mobile phone messages focused on blood pressure management reduce systolic blood pressure in adults with hypertension?
* Can FCHV home visits combined with regular mobile phone messages focused on diabetes management lower fasting blood glucose levels in adults with type 2 diabetes?
* Can FCHV home visits combined with regular mobile phone messages focused on smoking cessation increase the cessation rate among current smokers?

Researchers will compare the intervention group with a usual care group, which does not receive regular FCHV home visits for managing the three aforementioned risk factors or mobile phone messages.

DETAILED DESCRIPTION:
Background: Rapid globalization and urbanization continue to escalate the burden of non-communicable diseases (NCDs) across the world, disproportionally affecting low- and middle-income countries (LMICs). To date, trials have documented that task-sharing with community health workers (CHWs) can reduce systolic blood pressure and fasting blood glucose and achieve smoking cessation. However, most trials have been done in rural settings, and only focused on managing a single condition, such as hypertension. Furthermore, despite increasing evidence of the effectiveness from clinical trials, there is a lack of studies exploring best practices for 'how' to implement and sustain these interventions in LMICs.

Study Design: Type 2 hybrid effectiveness-implementation research study containing 1) a qualitative study, 2) open-label, two-armed, cluster randomized controlled trial (cRCT), and 3) implementation research plan. The details of the c-RCT only are presented below.

Settings: Pokhara Metropolitan City of Nepal. Pokhara is the second largest city in Nepal containing 33 administrative units called "wards". The investigators consider wards as clusters and randomize these 30 clusters (28 independent wards and 2 combined wards) into intervention and control groups in a 1:1 ratio.

Participants: Adults with ages between 40-75 having at least one of the following conditions:

* Hypertension, defined as:

  i. BP≥140/90 mmHg at two separate measures, or ii. Under pharmacotherapy for hypertension
* Type 2 diabetes mellitus, defined as i. Fingerprick glucose (fasting) ≥100 mg/dl, plasma glucose (fasting) ≥126 mg/dL, and ii. HbA1c ≥ 6.5 %, or iii. Under pharmacotherapies for type 2 diabetes
* Current tobacco smoking, defined as i. Ever smoked ≥100 cigarettes in lifetime, and ii. Currently smokes every day or on some days.

Intervention: Multifaceted intervention containing the following two components:

1. FCHV home visits every three months
2. Mobile phone messages, including

Control: Usual care in Pokhara Metropolitan City in Nepal, which does not include FCHV home visits for management of hypertension, diabetes, or smoking, and mobile phone messages.

Outcome: Changes in systolic blood pressure, fasting blood glucose, and smoking cessation at 6 months post randomization will be measured as primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting at least one of the following three conditions

   * Hypertensive, defined as
   * BP≥140/90 mmHg at two separate measurements
   * Type 2 diabetes, defined as
   * Fingerprick glucose≥100 mg/dL, and plasma fasting glucose ≥126 mg/dL, and HbA1c≥6.5
   * Current smoker, defined as
   * Ever smoked ≥100 cigarettes in lifetime, and
   * Currently smokes every day.
2. Registered on the voter list in Pokhara.
3. Not planning to migrate outside of Pokhara during the study period

Exclusion Criteria:

1. Blood pressure ≥180/120 mmHg or
2. Blood glucose >250 mg/dL or <54 mg/dL
3. Diagnosed with secondary hypertension by health professionals
4. Diagnosed with other diabetes besides type 2 by health professionals
5. Presenting with acute symptoms that may require hospitalizations, which includes but not limited to:

   * Nausea, vomiting, diarrhea
   * Abdominal pain
   * Polyuria, polydipsia, polyphagia
   * Loss of motor or sensory function
   * Altered mental status.
   * Chest pain, chest tightness
   * Dyspnea, shortness of breath
   * Fever
6. Diagnosed as terminally ill by a health professional, defined as life expectancy of 6 months or less.
7. Pregnant or intend to be pregnant

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2070 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (mmHg) | 6 months post randomization
  Difference in systolic blood pressure change between the intervention and the control groups among participants enrolled as having hypertension.
Fasting Plasma glucose | 6 months post randomization
  Difference in fasting plasma glucose change between the intervention and the control groups among participants enrolled as having type 2 diabetes.
Participants Who Have Achieved Smoking cessation | 6 months post randomization
  Participants who have not smoked for the past 30 days between the intervention and the control groups, among participants enrolled as current smokers.

SECONDARY OUTCOMES:
Diastolic blood pressure (mmHg) | 6 months post randomization
  Difference in diastolic blood pressure change between the intervention and the control groups among participants enrolled as having hypertension.
Controlled blood pressure control (<140/90 mmHg) rate | 6 months post randomization
  Difference in the proportion of those with BP<140/90 mmHg between the intervention and the control groups, among participants enrolled as having hypertension.
Mean HbA1c level | 6 months post randomization
  Difference in mean HbA1c between the intervention and the control groups, among participants enrolled as having type 2 diabetes.
Mean Weight in Kg | 6 months post randomization
  Difference in mean weight between the intervention and the control groups, among participants enrolled as having type 2 diabetes.
Mean Total Cholesterol (mg/dL) | 6 months post randomization
  Difference in mean total cholesterol levels between the intervention and the control groups, among participants with high total cholesterol (≥ 200 mg/dL) at baseline.
Mean HDL (mg/dL) | 6 months post randomization
  Difference in mean HDL levels between the intervention and the control groups, among participants with low HDL (< 40 mg/dL) at baseline.
Mean LDL level (mg/dL) | 6 months post randomization
  Difference in mean LDL levels between the intervention and the control groups, among participants with high LDL (≥ 100 mg/dL) at baseline.
Mean Triglyceride Levels (mg/dL) | 6 months post randomization
  Difference in mean triglyceride levels between the intervention and the control groups, among participants with high triglyceride level (≥ 150 mg/dL) at baseline.
Medication adherence, antihypertensive medicines | 6 months post randomization
  Difference in the proportion of those not missing a single anti-hypertensive pill over the past 1 week between the intervention and the control groups, among participants enrolled as having hypertension.
Medication adherence, hypoglycemic medicines | 6 months post randomization
  Difference in the proportion of those not missing a single hypoglycemic pill or injection over the past 1 week between the intervention and the control groups, among participants enrolled as having type 2 diabetes.
Fagerstrom Test for Nicotine Dependence (FTND) score | 6 months post randomization
  Difference in the proportion of those with a high FTND score (5-10) between the intervention and the control groups, among participants enrolled as current smokers. Higher means more dependence on nicotine.
Smoking cessation, 7 days | 6 months post randomization
  Difference in the proportion of those who have not smoked for the past 7 days between the intervention and the control groups, among participants enrolled as current smokers.
Harmful alcohol consumption rate, self-report | 6 months post randomization
  Difference in the proportion of those taking 7 (if women) and 14 (if men) standard drinks over the past 1 week between the intervention and the control groups, among all participants.
Low dietary salt intake rate, self-report | 6 months post randomization
  Difference in the proportion of those taking 5 mg or less salt per day between the intervention and the control groups, among participants enrolled as having hypertension.
High physical activity rate, self-report | 6 months post randomization
  Difference in the proportion of those who had 3000 metabolic equivalents of tasks (MET) or more per week between the intervention and control groups, among participants enrolled as having hypertension and/or diabetes.
High fruit and vegetable intake rate, self-report | 6 months post randomization
  Difference in the proportion of those who consumed 5 or more servings of fruits and/or vegetables per day between the intervention and control groups, among participants enrolled as having hypertension and/or diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Neupane, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Pokhara Metropolitan City, Pokhara, Gandaki, Nepal

IPD SHARING:
Plan to Share IPD: No